CLINICAL TRIAL: NCT00428688
Title: Assessment of Endothelial Function and IMT in Survivors Hodgkin's Lymphoma Patients
Brief Title: Endothelial Function and IMT in Survivors of Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Dalit Modan, Pediatirc Endocrinologist, Sheba Medical Center
Other Study IDs: SHEBA-06-4359-DM-CTIL
Record Dates: First submitted 2007-01-28; First posted 2007-01-30 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's lymphoma; cardiovascular disease; radiation therapy; Brachial artery flow-mediated dilation (FMD)
MeSH Terms: conditions — Hodgkin Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the proposed study is to assess endothelial function and IMT, as correlates of cardiovascular disease (CVD), in young adult Hodgkin's disease (HD) survivors, and to relate endothelial function to other risk factors including obesity, dyslipidemia, hyperinsulinemia and fasting glucose.

DETAILED DESCRIPTION:
Disease free survival of Hodgkin's disease (HD) patients has improved dramatically over the past few decades. With the dramatic advance in patient's survival, the prevention and treatment of long-term adverse effects of chemotherapy and radiotherapy has become a major focus of interest. HD survivors have excess mortality compared with the age-matched general population, even after excluding disease relapse. A considerable proportion of the excess mortality is due to cardiovascular disease (CVD), principally ischemic heart disease and stroke.

The proposed study will assess endothelial function in HD survivors, using the non-invasive technique of brachial artery flow-mediated dilation (FMD), by high-resolution ultrasonography. We will also assess IMT. The results of these tests are independent predictors of atherosclerosis disease progression and cardiovascular event rates. This is a prospective study comprising 40 young-adult (aged 18-30 years) . The study will comprise 40 survivors of HD: 20 patients treated with chemotherapy and radiotherapy to the chest and 20 patients treated with chemotherapy alone. The patients will be compared to age and sex-matched patients from the data base of the endothelial function laboratory at the heart institute of the Sheba Medical Center. In addition to brachial artery endothelial function assessment, the patients will also undergo a physical examination including anthropometric measurements (height, weight, waist and hip circumference), and blood pressure. The evaluation will also include blood tests for glucose, lipid profile, CRP, AST, ALT and insulin. A medical history including smoking history and family history of CVD and dyslipidemia will be obtained.

Patients treated with radiotherapy to the chest will be compared to patients treated with chemotherapy alone and both patients will be compared to healthy controls. The patients will be characterized by age, risk factors for coronary heart disease and endothelial function as assessed by brachial artery FMD. We will establish the rate of endothelial function abnormalities in survivors of HD and its correlation with the other risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin's disease survivors over 18 years old

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young-adult survivors of Hodgkin's disease
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Frequencey of endothelial dysfunction by FMD | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dalit Modan, M.D, Principal Investigator — Sheba Medical Center; Michael Schechter, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- The Endothelaial function lab, The Heart Institute, Sheba Medical Center, Israel, Ramat Gan, Israel